CLINICAL TRIAL: NCT05681143
Title: A Crisis Prevention Program in Youth With Autism Spectrum Disorder
Brief Title: A Crisis Prevention Program for Youth With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00332878
Record Dates: First submitted 2022-12-30; First posted 2023-01-12 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder; Behavior Problem
Keywords: autism; externalizing; behavior; crisis
MeSH Terms: conditions — Autism Spectrum Disorder; Mental Disorders; Autistic Disorder; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crisis Prevention Arm (Active Comparator)
  Interventions: Other: Crisis Prevention Arm
- Control (Placebo Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Crisis Prevention Arm — The crisis prevention program involves a 3-session model. Each session lasts up to 60 minutes. They take place via telehealth with a licensed clinical therapist. Sessions involve case formulation, provision of prevention strategies, connecting with professional and lay resources, what to do if a crisis occurs, and strategies to prevent the re-occurrence of a crisis, should one occur. Each session involves use of checklists, a community resource guide, and homework. Implementation is standardized using two different manuals, one for the parent and the other for the provider.
  Arms: Crisis Prevention Arm
Other: Control — The control condition will involve sending families the Autism Speaks Challenging Behavior Toolkit. It offers a complimentary set of recommendations. It is freely available and can be found here: https://www.autismspeaks.org/tool-kit/challenging-behaviors-tool-kit. There is no interaction with the clinician in the controlcondition. After the study observation period, we will provide them with the crisis manual (for parents) used in the active treatment arm.
  Arms: Control

SUMMARY:
Mental health crises involve acute psychiatric states, such as aggression and/or self-injury, which can result in harm to self or others. There is evidence to suggest that 20% to 25% of autistic children are at risk of a mental health crises, however no crisis prevention programs exist for autistic children. The goal of this project is to evaluate, via a randomized design, a novel crisis prevention program.

DETAILED DESCRIPTION:
When a child or adolescent experiences a mental health crisis, it is a devastating and potentially life-threating event. Beyond the hazard of injury, mental health crises can have a life-altering impact on the child (repeated trauma, development of future psychopathology), family members (increased stress and poorer well-being) and society as a whole (cost and disability). Our inability to prevent or identify those in crisis is reflected in the rising rates of suicides, extensive wait times and overcrowding in emergency departments, and the jailing of people with mental illness.

Mental health crises are defined as a) the presence of acute psychiatric symptoms that require immediate attention or intervention and b) the perceived (by the informant) lack of immediate resources to manage these symptoms. Similar to the concepts of impairment or distress, mental health crisis is a transdiagnostic construct that applies to all psychiatric problems, from self-injury to aggression to psychosis to substance abuse.

The recently developed Mental Health Crisis Assessment Scale-Revised (MCAS-R), developed by a team of expert clinical and public health researchers, was specifically designed to address the current gap in crisis measurement for autistic children. The MCAS-R is a 23-item parental report, which takes no more than 10 minutes to complete, that measures crisis in two conceptually-based subscales, acuity and behavioral efficacy, reflecting both the core elements of crisis. Based on the cutoffs, it has been shown to accurately identify crises in 9 out of 10 autistic children. Recent work suggests between 20-25% of children served in outpatient mental health are at risk of a mental health crisis, as identified by the validated MCAS cutoff.

At present, no crisis prevention programs exist for autistic children. There are certainly numerous community-based crisis intervention programs, outpatient mental health treatment approaches, and parent behavioral training programs. However, no programs exist that aim to prevent a crisis from occurring. The goal of this study is to fill this gap by providing families with tools before their child's behavior becomes acute.

The goals of this study are to examine: 1) child and parent outcomes associated with a novel crisis prevention program for autistic children; 2) gather survey-based feedback from parents, post-intervention, to understand feasibility and utility of the crisis prevention program.

ELIGIBILITY:
Inclusion Criteria:

* Have a child with autism
* The child must be 3-17 years of age
* Caregivers must score <=13 on the Crisis Prevention Index (CPI)
* The child must have some behavioral concerns (e.g., aggression, property destruction, elopement, tantrums), as listed on section 2 of the MCAS-R.
* The child must have an MCAS-R Acuity score of at most 19
* The child must be actively seen by a medical or mental health professional within the last six months

Exclusion Criteria:

* The child has any suicidal thoughts or behaviors
* The child is enrolled in another treatment study
* The child is enrolled in the RUBI parent training program, offered at the Center for Autism and Related Disorders at Kennedy Krieger
* Caregivers has a hearing or language impairment
* Caregiver does not have consistent access to the internet

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Change in The Crisis Prevention Index scores | baseline, 4 weeks, 8 weeks
  5-item, custom measure assessing caregivers perceived preparation for a crisis involving their child. Higher scores are better.

SECONDARY OUTCOMES:
Change in Me as a Parent Scale scores | baseline, 4 weeks, 8 weeks
  16-item measure assessing caregivers perceived ability to manage their child's behavior. Higher scores are better.
Change in Mental Health Crisis Assessment Scale-Revised scores | baseline, 4 weeks, 8 weeks
  23-item parental report that measures crisis in two conceptually-based subscales, acuity and behavioral efficacy, reflecting both the core elements of crisis. Higher scores are worse.
Change in Aberrant Behavior Checklist scores | baseline, 4 weeks, 8 weeks
  58-item measure of child behavior problems. Higher scores are worse.

CONTACTS AND LOCATIONS:
Overall Officials: Luther Kalb, PhD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vasa RA, Hagopian L, Kalb LG. Investigating mental health crisis in youth with autism spectrum disorder. Autism Res. 2020 Jan;13(1):112-121. doi: 10.1002/aur.2224. Epub 2019 Oct 25. PMID 31652032
- [Background] Kalb LG, DiBella F, Jang YS, Fueyo M, Mahajan R, Vasa RA. Mental Health Crisis Screening in Youth with Autism Spectrum Disorder. J Clin Child Adolesc Psychol. 2025 Jan-Feb;54(1):127-135. doi: 10.1080/15374416.2022.2119984. Epub 2022 Sep 21. PMID 36129785